CLINICAL TRIAL: NCT03403647
Title: The Effect of Normalizing Vitamin D Concentrations on Everlomius Trough Concentrations
Brief Title: Effect of Vitamin D on Everolimus Trough Concentrations Among Heart Transplanted Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sheba Medical Center (Other Government)
Responsible Party: Principal Investigator, Dr.Itai Gueta, Physician in the institute for clinical pharmacology, Sheba Medical Center
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Vitamin D and Everolimus
Record Dates: First submitted 2018-01-11; First posted 2018-01-18 (Actual); Last update posted 2019-04-18 (Actual); Status verified 2019-04

CONDITIONS: Vitamin D Deficiency
MeSH Terms: conditions — Vitamin D Deficiency | interventions — Vitamin D

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Vitamin D deficient (Experimental): Vitamin D supplementation and close everolimus trough levels monitoring with oral dose adjustments
  Interventions: Dietary Supplement: Vitamin D
- No vitamin D deficiency (No Intervention): Regular and routine monitoring

INTERVENTIONS:
Dietary Supplement: Vitamin D — Oral daily vitamin D
  Arms: Vitamin D deficient

SUMMARY:
Vitamin D is part of the regular treatment regimen among patients after heart transplantation. Due to potential drug-drug interaction between vitamin D and everolmus, these patients are in increased risk for increased everolimus metabolism, potentially leading to under- immunosupression.

DETAILED DESCRIPTION:
post heart transplantation patients treated with everolimus will be screened for vitamin D levels. Patients defined as deficient will be treated with vitamin D with close and intensive monitoring everolimus levels, adjusting oral daily dose to maintain therapeutic levels.

ELIGIBILITY:
Inclusion Criteria:

Heart transplanted patients treated with everolimus

Exclusion Criteria:

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2018-07-15 (Actual); Primary Completion 2019-04-10 (Actual); Study Completion 2019-04-10 (Actual)

PRIMARY OUTCOMES:
Oral daily everolimus dose change | 8 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Sheba Medical Center, Ramat Gan, Israel